CLINICAL TRIAL: NCT00757887
Title: Re-exposure of EHMI-8 Human Volunteers to Live Malaria Sporozoites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Prof. Dr. R.W. Sauerwein, Radboud University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EHMI-8B
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2009-10

CONDITIONS: P. Falciparum Malaria
Keywords: malaria; plasmodium; falciparum; human; experimental infection
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EHMI8 (Experimental): Previously protected volunteers, N=10
  Interventions: Biological: Exposure to 5 P. falciparum infected mosquitoes
- control (Active Comparator): 5 malaria-naive volunteers
  Interventions: Biological: Exposure to 5 P. falciparum infected mosquitoes

INTERVENTIONS:
Biological: Exposure to 5 P. falciparum infected mosquitoes — Five Anopheles Stephensi mosquitoes are infected with NF54 P.falciparum. volunteers are exposed to bites for 10 minutes.

SUMMARY:
In the EHMI-8 study (CMO 2006/207) the investigators induced sterile protection against P. falciparum challenge in healthy Dutch volunteers by repeated exposure to infected mosquitoes whilst under chloroquine prophylaxis. The surprisingly efficient induction of protection in this study strongly supports the development of whole parasite vaccines and is therefore an important finding to malaria vaccine development. In this study (EHMI8B) the investigators would like to explore the longevity of the protective immune response and simultaneously further characterise immune mechanisms responsible for protection by re-exposing EHMI-8 volunteers to infected mosquito bites.

ELIGIBILITY:
Inclusion criteria

1. Age > 18 and < 35 years healthy volunteers (males or females).
2. General good health based on history and clinical examination.
3. Negative pregnancy test.
4. Use of adequate contraception for females
5. All volunteers have to sign the informed consent form following proper understanding of the meaning and procedures of the study
6. Volunteer agrees to inform the general practitioner and agrees to sign a request for medical information concerning contra-indications for participation in the study
7. Willingness to undergo a P. falciparum sporozoite challenge
8. Resident near the RUNMC, Nijmegen or agree to stay in a hotel room during the intensive period of the study (Day 5 till Day T +3)
9. Reachable by mobile phone during the whole study period
10. Availability to attend all study visits
11. Agreement to refrain from blood donation to Sanquin or for other purposes, during the course of the study
12. Willingness to undergo an HIV, hepatitis B and C test
13. Negative urine toxicology screening test at screening visit and day before challenge

Exclusion criteria

1. History of malaria other than participation in EHMI-8, or residence in malaria endemic areas within the past six months
2. Plans to travel to endemic malaria areas during the study period.
3. Only for newly recruited control volunteers: previous participation in any malaria vaccine study and/or positive serology for P. falciparum
4. Symptoms, physical signs and laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers.
5. History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
6. History of arrhythmia's or prolonged QT-interval
7. Positive family history in 1st and 2nd degree relatives of cardiac disease < 50 years old
8. An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.
9. Any clinically significant deviation from the normal range in biochemistry or haematology blood tests or in urine analysis
10. Positive HIV, HBV or HCV tests
11. Participation in any other clinical study within 30 days prior to the onset of the study
12. Volunteers enrolled in any other clinical study during the study period
13. Pregnant or lactating women
14. Volunteers unable to give written informed consent
15. Volunteers unable to be closely followed for social, geographic or psychological reasons
16. Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
17. A history of psychiatric disease
18. Known hypersensitivity for anti-malaria drugs
19. History of severe reactions or allergy to mosquito bites
20. The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months before study onset (inhaled and topical corticosteroids are allowed) and during the study period
21. Contra-indications to Malarone® including treatment taken by the volunteers that interfere with Malarone®
22. Any confirmed or suspected immunosuppressive or immunodeficiency condition, including asplenia
23. Co-workers of the departments of Medical Microbiology or Internal Medicine of the Radboud University Nijmegen Medical Centre

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
A significant difference in time of thick smear positivity between EHMI-8 and control volunteers | 21 days
A significant quantitative difference in parasitemia as measured by PCR between EHMI-8 and control volunteers | 21 days
A significant difference in kinetics of parasitemia between EHMI-8 and control volunteers as measured by PCR. | 21 days
A difference in occurrence of signs or symptoms between EHMI-8 and control volunteers | 21 days

SECONDARY OUTCOMES:
Difference in immunological parameters between EHMI-8 and control volunteers. | 140 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- UMC St. Radboud, Nijmegen, Netherlands

REFERENCES:
- [Derived] Coffeng LE, Hermsen CC, Sauerwein RW, de Vlas SJ. The Power of Malaria Vaccine Trials Using Controlled Human Malaria Infection. PLoS Comput Biol. 2017 Jan 12;13(1):e1005255. doi: 10.1371/journal.pcbi.1005255. eCollection 2017 Jan. PMID 28081133
- [Derived] Roestenberg M, Teirlinck AC, McCall MB, Teelen K, Makamdop KN, Wiersma J, Arens T, Beckers P, van Gemert G, van de Vegte-Bolmer M, van der Ven AJ, Luty AJ, Hermsen CC, Sauerwein RW. Long-term protection against malaria after experimental sporozoite inoculation: an open-label follow-up study. Lancet. 2011 May 21;377(9779):1770-6. doi: 10.1016/S0140-6736(11)60360-7. Epub 2011 Apr 22. PMID 21514658